CLINICAL TRIAL: NCT04786405
Title: An Experimental, Randomized Trial Comparing Mindfulness Meditation Versus Clinical Hypnosis for Acute Pain: a Test of Effects and Mechanisms
Brief Title: Mindfulness Meditation Versus Clinical Hypnosis for Acute, Experimental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #2019000347
Record Dates: First submitted 2021-02-28; First posted 2021-03-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Mindfulness Meditation; Clinical Hypnosis
Keywords: Mindfulness Meditation; Hypnosis; Acute Pain; Experimental Pain; Mechanisms
MeSH Terms: conditions — Acute Pain | interventions — Mindfulness; Hypnosis

STUDY DESIGN:
Intervention Model Description: Single-blind, two-arm, parallel-group randomized design.
Who Masked: Outcomes Assessor
Masking Description: The experimenter will remain blind to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation (Experimental): Participants in this arm will complete five, 20-minute mindfulness meditation sessions delivered over consecutive days.
  Interventions: Behavioral: Mindfulness meditation
- Clinical Hypnosis (Active Comparator): Participants in this arm will complete five, 20-minute clinical hypnosis sessions delivered over consecutive days.
  Interventions: Behavioral: Clinical hypnosis

INTERVENTIONS:
Behavioral: Mindfulness meditation — Participants in the mindfulness meditation condition will practice a breath and body focused meditation.
  Arms: Mindfulness Meditation
Behavioral: Clinical hypnosis — Participants in clinical hypnosis will be guided in a hypnosis practice with suggestions tailored towards shifting pain appraisals.
  Arms: Clinical Hypnosis

SUMMARY:
This trial aims to determine the effects and mechanisms (mediators and moderators) of brief training in mindfulness meditation versus clinical hypnosis on acute, experimental pain.

DETAILED DESCRIPTION:
Participants (N=200 with complete data) will be healthy undergraduate students or community-based individuals. An experimental, randomised trial will be implemented, with participants randomly assigned to either five daily, 20-minute mindfulness meditation sessions or clinical hypnosis sessions. Repeated measures and experimental pain manipulation will be implemented. Aim 1 is to examine the effects of these two treatments on experimental pain outcomes. Aim 2 is to examine the moderators of these effects. Aim 3 is to determine the mediators underlying improved experimental pain outcomes. Results will refine theory and will inform the future streamlining of treatments to target those mechanisms shown to be of most critical importance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Able to read, speak and understand English.

Exclusion Criteria:

* Pregnancy, heart or vascular disease, Raynaud's disease, sickle cell disease, seizure disorder, high blood pressure, or diabetes;
* Experience of recurrent fainting spells;
* Report of a chronic pain condition;
* Use of alcohol and/or pain medication in the last 24-hours;
* Currently receiving psychiatric care;
* Problems with allergic skin reactions or excessive bruising;
* Previous participation in a cold pressor experiment.
* All participants will be asked to consume a fruit box drink prior to the cold pressor to prevent vasovagal reactions.

These exclusion criteria are standard when using a cold pressor task in a healthy undergraduate population and ensure safe procedures to mitigate any potential risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Pain unpleasantness | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  Numerical rating scale in response to exposure to a cold pressor task.
Pain intensity | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  Numerical rating scale in response to exposure to a cold pressor task.
Pain tolerance | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  How long (in seconds) participants tolerate the cold pressor task with the time starting at the point of immersion and stopping when the hand, wrist and forearm were withdrawn from the refrigerated water.

SECONDARY OUTCOMES:
Physiological response to pain stimulus | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  Heart rate data
Mechanism: Attention Network Task | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  A computer based task that has been developed to allow assessment of the functioning of the three major attentional networks; alerting, orienting, and executive attention.
Mechanism: Mind Wandering Task | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  A computer based task that has been developed to allow assessment of three types of mind wandering.
Mechanism: Mindfulness | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  Five Facet Mindfulness Questionnaire-Short Form
Mechanism: Pain catastrophizing | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  Pain Catastrophizing Scale
Mechanism: Pain appraisals | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  Pain Appraisal Inventory
Mechanism: Pain-Related Cognitive Processes | Change from Experimental Session 1 (Day 1) to Experimental Session 5 (Day 5)
  Pain-Related Cognitive Process Questionnaire34
Mechanism: Hypnotizability | Baseline score at Experimental Session 1 (Day 1)
  Stanford Clinical Hypnotizability Scale
Mechanism: Pre-treatment expectancies | Baseline score at Experimental Session 1 (Day 1)
  Treatment Expectations Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
We will make available to interested researchers a data file containing the de-identified data used for each published article at the time that the article is accepted for publication. The data will be de-identified to remove any variables from which it would be possible to identify any individual participants. Specifically, we will create a data file that includes all of the variables used in any published article and a list of the variables in the data file (along with their variable labels) and email to investigators who request the data a copy of: (1) the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) a copy of the data set (as an SPSS.sav file).